CLINICAL TRIAL: NCT05703477
Title: The Dynamic Fluctuation of Donor Microbiota Affects the Prognosis of Fecal Microbiota Transplantation for C. Difficile Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Shanghai Tenth People's Hospital, Tenth People's Hospital of Tongji University, Shanghai 10th People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMTCDI
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Clostridium Difficile Infection; Fecal Microbiota Transplantation
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT Responder (Experimental)
  Interventions: Procedure: Fecal microbiota transplantation
- FMT non-Responder (Experimental)
  Interventions: Procedure: Fecal microbiota transplantation

INTERVENTIONS:
Procedure: Fecal microbiota transplantation — Fecal microbiota transplantation (FMT) achieves the purpose of treating intestinal and extra-intestinal diseases by transplanting the functional microbes in the feces of healthy people into the patient's intestine through the upper or lower alimentary tract routes to rebuild the patient's intestinal microbiota.

SUMMARY:
Fecal microbiota transplantation (FMT) achieves the purpose of treating intestinal and extra-intestinal diseases by transplanting the functional microbes in the feces of healthy people into the patient's intestine through the upper or lower alimentary tract routes to rebuild the patient's intestinal microbiota. Recently, FMT has been widely used in the treatment of various gastrointestinal diseases, including but not limit in CDI. In this study, we focused on the demonstration of FMT action mechanism in CDI treatment.

ELIGIBILITY:
Inclusion Criteria:

1. aged over 18 years old;
2. positive stool test for Clostridium difficile 16S rDNA and/or glutamate dehydrogenase;
3. can tolerate nasojejunal tube and complete full course of FMT treatment;
4. the clinical data are relatively complete and there is follow-up available for evaluation

Exclusion Criteria:

1. accompanied by chronic wasting diseases such as malignant tumor and hyperthyroidism;
2. associated with gastrointestinal organic diseases such as short bowel syndrome, intestinal fistula, and inflammatory bowel disease; c) severe destruction of the intestinal mucosa, severe immunosuppression, combined with severe systemic infection; d) Intervention with antibiotics during treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
changes of microbiota before and after FMT treatment | 7 days, 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Hongliang Tian, Principal Investigator — Intestinal Microenvironment Treatment Center of General Surgery, Shanghai Tenth People's Hospital, Tenth People's Hospital of Tongji University
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided